CLINICAL TRIAL: NCT00057733
Title: Stress Management Training For Patients Undergoing Radiotherapy
Brief Title: Stress Management Training in Patients Undergoing Radiation Therapy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: MCC-0108; CDR0000069466 (Registry Identifier: PDQ (Physician Data Query)); NCI-5721; NCI-P02-0227; TAGH-20291
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-04

CONDITIONS: Anxiety Disorder; Depression; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: anxiety disorder; depression; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Stress management techniques such as muscle relaxation, guided imagery, and abdominal breathing may improve quality of life and decrease emotional distress in patients who are undergoing radiation therapy for cancer.

PURPOSE: Randomized clinical trial to determine the effectiveness of stress management training in helping cancer patients cope with the emotional distress of radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether a modified version of a self-administered stress management training intervention, previously found to be of benefit in chemotherapy patients, is effective in improving quality of life and decreasing psychological distress (anxiety and depression) in patients with cancer who are undergoing radiotherapy.

Secondary

* Compare the efficacy of this intervention on improving quality of life and decreasing psychological distress (anxiety and depression) in male vs female patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive self-administered stress management training (SSMT) in 3 stress management techniques (progressive muscle relaxation training and guided imagery, abdominal breathing, and coping skills) adapted specifically for use during radiotherapy. Patients initially receive a 5-minute standardized presentation regarding the nature and purpose of SSMT. Patients then receive information and instruction regarding the three stress management techniques comprising a videotape, audiotape, and brochure. Patients also receive their institution's usual psychosocial care.
* Arm II: Patients receive their institution's usual psychosocial care only. Quality of life, anxiety, and depression are assessed at baseline and then at 1, 2, and 3 weeks. Intervention helpfulness is assessed at 3 weeks.

PROJECTED ACCRUAL: A total of 327 patients (approximately 163 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Must be scheduled to receive a minimum of 12 radiotherapy treatments over a 21-day period

  * Must not be scheduled to receive CNS irradiation
  * Must not be scheduled to receive radiotherapy as palliative care only
  * Prostate seed implants allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to read and speak English

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy
* No concurrent cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2005-04 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Jacobsen, PhD, Study Chair — University of South Florida
Locations (12):
- United States (12):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Howard University Cancer Center at Howard University Hospital, Washington D.C., District of Columbia
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Comprehensive Cancer Care Center at Bethesda Memorial Hospital, Boynton Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Cancer Care and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Northwest, Tacoma, Washington